CLINICAL TRIAL: NCT03604848
Title: GRACE-TB：NGS-guided Regimens of Anti-tuberculosis Drugs for the Control and Eradication of MDR-TB
Brief Title: NGS-Guided(G) Regimens(R) of Anti-tuberculosis(A) Drugs for the Control(C) and Eradication(E) of MDR-TB
Acronym: GRACE-TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2018-291
Record Dates: First submitted 2018-06-26; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Multidrug Resistant Tuberculosis; next generation sequencing; drug susceptibility test; precision treatment
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NGS-guided regimen: Regimen A (Experimental): Regimen A: 9-month regimen for simple MDR-TB patients 4 months of pyrazinamide, amikacin ,moxifloxacin, prothionamide, and cycloserine , followed by 5months of pyrazinamide,moxifloxacin, prothionamide, and cycloserine
  Interventions: Drug: NGS-guided regimen: Regimen A
- NGS-guided regimen: Regimen B (Experimental): Regimen B: 12-month simple MDR-TB regimen for simple MDR-TB patients 6 months of pyrazinamide, amikacin ,moxifloxacin, prothionamide, and cycloserine , followed by 6 months of pyrazinamide,moxifloxacin, prothionamide, and cycloserine
  Interventions: Drug: NGS-guided regimen: Regimen B
- NGS-guided regimen: Regimen C (Experimental): Regimen C : for complicated MDR-TB patients In regimen C, the resistant drug(s) will be replaced by the other WHO recommended drugs for MDR-TB such as linezolid, clofazimine or ethambutol based on the drug susceptibility test results. The duration of treatment in the "complicated MDR-TB group" is consistent with control group, with 6 months of intensive phase and 18 months of consolidation phase.
  Interventions: Drug: NGS-guided regimen: Regimen C
- WHO-approved MDR-TB regimen (Active Comparator): 6 months of pyrazinamide, amikacin,moxifloxacin, prothionamide , and cycloserine , followed by 18 months of pyrazinamide, moxifloxacin, prothionamide , and cycloserine
  Interventions: Drug: WHO-approved MDR-TB regimen

INTERVENTIONS:
Drug: WHO-approved MDR-TB regimen — Pyrazinamide 33-50kg 1000-1750 mg daily, 51-70kg 1750-2000 daily, >70kg 2000-2500mg daily; Amikacin 600mg daily ; Moxifloxacin 33-50kg 400 mg daily, 51-70kg 600mg daily, >70kg 800mg daily; Prothionamide 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily ; Cycloserine 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily All treatment is taken daily.
  Arms: WHO-approved MDR-TB regimen
Drug: NGS-guided regimen: Regimen A — Pyrazinamide 33-50kg 1000-1750 mg daily, 51-70kg 1750-2000 daily, >70kg 2000-2500mg daily; Amikacin 600mg daily ; Moxifloxacin 33-50kg 400 mg daily, 51-70kg 600mg daily, >70kg 800mg daily; Prothionamide 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily ; Cycloserine 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily All treatment is taken daily.
  Arms: NGS-guided regimen: Regimen A
Drug: NGS-guided regimen: Regimen B — Pyrazinamide 33-50kg 1000-1750 mg daily, 51-70kg 1750-2000 daily, >70kg 2000-2500mg daily; Amikacin 600mg daily ; Moxifloxacin 33-50kg 400 mg daily, 51-70kg 600mg daily, >70kg 800mg daily; Prothionamide 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily ; Cycloserine 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily All treatment is taken daily.
  Arms: NGS-guided regimen: Regimen B
Drug: NGS-guided regimen: Regimen C — Based on the drug susceptibility test results, the resistant drug(s) will be replaced by the other WHO recommended drugs for MDR-TB such as linezolid, clofazimine or ethambutol.
  The dose of linezolid, clofazimine or ethambutol as follows:
  Linezolid: 600 mg daily, clofazamine: 33-50kg 50 mg daily, 51-70kg 100 daily, >70kg 100 mg daily; ethambutol: 33-50kg 800 mg daily, 51-70kg 800 daily, >70kg 1200 mg daily;
  Arms: NGS-guided regimen: Regimen C

SUMMARY:
Tuberculosis (TB) has been one of the top 10 causes of death worldwide from a single infectious agent, ranking above HIV/AIDS. Management and eradication of this disease is being hindered by the emergence of multidrug-resistant TB (MDR-TB) and extensively drug resistant TB (XDR-TB). Globally, there were estimated 10.4 million cases of TB and 490,000 cases of MDR-TB in 2016. China accounts for around 8.6% (0.895/10.4 million) of the global TB burden, ranking third in the top 3 countries (India, Indonesia, China) with the highest number of TB cases and ranking first with the largest number of MDR/ Rifampin-Resistant (RR)-TB cases. The treatment success rate for MDR-TB using the 18-24-month conventional World Health Organization (WHO) regimen was estimated to be about 54% worldwide and 41% for China in 2016, which remains unacceptably low.

The poor MDR-TB treatment success rates suggest that current drug regimens are suboptimal. In addition, they are costly with a high pill burden, as many drugs, with significant potential for adverse events, are given for a long duration. These factors also inhibit good treatment compliance with further negative impact on treatment outcomes. According to previous studies, treatment outcomes of MDR-TB could be affected by drug resistance of pivotal drugs in MDR-TB regimen, such as fluoroquinolones, second-line injectable agents and pyrazinamide. The available drug-resistance information could help physicians decide the proper regimens for MDR-TB patients, which may prevent the useless prescription and evitable adverse.

Therefore, the individualized regimen based on the resistance profile of the bacteria and patients' drug tolerance should be aimed for high-quality treatment for MDR-TB in the future. A precision individualized treatment approach based on the rapid molecular drug susceptibility tests of second line drugs may assist clinicians in making more suitable regimen and improve the treatment outcome of MDR-TB. Also, precision regimen offers the opportunity to improve treatment of drug-resistant tuberculosis through reduced toxicity while reducing the risk of resistance amplification and further transmission at a population level.

The purpose of this research is to assess the feasibility and effects of individualized regimen that is guided by rapid molecular drug susceptibility tests of key second-line drugs through next generation sequencing. Meanwhile, the study will evaluate a short course regimens of drugs among "simple MDR-TB" patients who are proven to be sensitive to fluoroquinolones ,injectable second-line drugs and pyrazinamide.

DETAILED DESCRIPTION:
The GRACE-TB study is a multi-center, open-label, randomized, controlled trial in patients with MDR-TB. This study will assess the feasibility and effects of individualized regimen for MDR-TB based on rapid molecular drug susceptibility tests（DSTs） of key second-line drugs through next generation sequencing (NGS) and try to improve the treatment outcome of MDR-TB. And the study will evaluate a shorter course regimen among patients who are proven to be sensitive to fluoroquinolones (FQs) or second-line injectable drugs(SLIDs) or pyrazinamide (PZA) through NGS.

A total of 488 participants with MDR-TB will be recruited and followed up until 18 months after the end of treatment. During randomization, eligible patients will be assigned in a 1:3 ratio to one of the following groups: a control group, which is treated with WHO-approved MDR-TB regimen, composed of 6 months of PZA, amikacin (Am) ,moxifloxacin (MFX), prothionamide (PTO), and Cycloserine (Cs), followed by 18 months of PZA, MFX, PTO and Cs; a NGS-guided group, which is treated with one individualized regimen that is guided by the drug susceptability test results of FQs/PZA/ SLIDs through NGS.

About 366 patients will be enrolled in the NGS-guided group. Based on the molecular DST results of FQs/PZA/ SLIDs , patients proven to be sensitive to PZA, FQs and SLIDs will be divided into to the "simple MDR-TB group" and those with resistant to at least one of FQs/PZA/ SLIDs will be divided into to "complicated MDR-TB group".

Patients in the "simple MDR-TB group" will be assigned randomly in a 1:1 ratio to one of the following daily regimen: a 9-month regimen(Regimen A) which consists of 4-month intensive therapy of PZA, Am, MFX,PTO, Cs, followed by 5-month consolidation therapy of PZA, MFX, PTO and Cs; a 12-month regimen(Regimen B) which consists of 6-month intensive therapy of PZA, Am, MFX,PTO, Cs, followed by 6-month consolidation therapy of PZA, MFX, PTO and Cs.

Patients in the "complicated MDR-TB group" will be treated a regimen (Regimen C) in which the resistant drug(s) will be replaced by the other WHO recommended drugs for MDR-TB such as linezolid, clofazimine or ethambutol based on the DST results. The duration of treatment in the "complicated MDR-TB group" is consistent with control group, with 6 months of intensive phase and 18 months of consolidation phase.

The primary objective is to compare the proportion of patients with a favorable efficacy between the NGS-guided group and the control group. The second objective is to assess whether the proportion of simple MDR-TB patients with a favorable efficacy outcome of Regimen A is not inferior to Regimen B. The participants will be followed up to 18 months after the end of the treatment. The data accrued to 18 months after the end of treatment will be used in primary and secondary analyses.

Safety evaluations performed are the routine lab tests, blood glucose, hearing, vital signs, electrocardiograph (ECG), reporting of adverse events, physical examinations and chest CT. Adverse events will be monitored and promptly managed during the whole treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with active MDR-TB. MDR-TB is defined as resistance to the following two drugs: Isoniazid and Rifampicin.
* Patients who are smear positive and sputum culture positive for mycobacterium tuberculosis
* HIV negative.
* The patients should be voluntarily entering the study and willing to sign up the consent form after full knowledge of the risks, schedule, drug features of this study.

Exclusion Criteria:

* Known allergy or intolerance to the drugs in this study
* Liver damage (Hepatic encephalopathy; ascites; prothrombin time prolonged 2 seconds compared with normal controls; blood bilirubin 3 times greater than the upper limit of the normal range)
* Platelets <150x10^9 / L, WBC < 3x10^9 / L.
* Abnormal ECG (Male patients with prolonged QT interval exceeding 430ms,
* Female patients with prolonged QT interval exceeding 450ms)
* Serum creatinine 1.5 times higher than upper limit
* Fasting blood-glucose higher than 8.0 mmol/L
* Patients who are on medication that effect the results of the drugs in this study Karnofsky score<50% (see appendix)
* Women who are pregnant or breastfeeding
* HIV positive
* Participating in other clinical trials in the past three months
* Patients with mental illness and severe neurosis
* Patients who have poor compliances
* Any special circumstances in which the research physicians believe that is not suitable for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2018-08-05 (Estimated); Primary Completion 2024-08-04 (Estimated); Study Completion 2024-08-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NGS-guided treatment(the proportion of patients with a favorable efficacy outcome 18 months after the end of treatment) | 18 months after the end of treatment
  to compare the proportion of patients with a favorable efficacy outcome between the NGS-guided group and conventional WHO-approved MDR-TB group

SECONDARY OUTCOMES:
Efficacy of shorter course regimen for simple MDR-TB patients(the proportion of patients with a favorable efficacy outcome between regimen A and regimen B) | 18 months after the end of treatment
  to assess whether the proportion of simple MDR-TB patients with a favorable efficacy outcome of Regimen A is not inferior to Regimen B
Safety(the proportion of patients who experience grade 3 or greater adverse events) | 18 months after the end of treatment
  to compare the proportion of patients who experience grade 3 or greater adverse events (graded according to the Division of AIDS severity criteria for adverse events), during treatment or follow-up, on the experimental regimen when compared to the control regimen;
The Median Time to Sputum Culture Conversion | 24 months after the start of treatment
  time from treatment initiation to the first of two consecutive negative sputum cultures without an intervening positive culture in liquid media between the NGS-guided group and conventional WHO-approved MDR-TB group;

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD,MD, Principal Investigator — Huashan Hospital of Fudan University, Shanghai, China
Locations (12):
- China (12):
  - The Third People's Hospital of Shenzhen City, Shenzhen, Guangzhou
  - the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Chest Hospitalof Xinjiang Uygur Autonomous Region of PRC, Ürümqi, Xinjiang
  - Zhuji City People's Hospital, Zhuji, Zhejaing
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang
  - The Second Hospital of Yinzhou of Ningbo, Ningbo, Zhejiang
  - Enze Medical Center of Taizhou CIty, Taizhou, Zhejiang
  - The Central Hospital of Wenzhou City, Wenzhou, Zhejiang